CLINICAL TRIAL: NCT02977910
Title: Comparative Study for Ankle Fracture Combined With Deltoid Ligament Rupture
Brief Title: Treatment Strategy of Ankle Fracture Combined With Deltoid Ligament Rupture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liming Cheng (Other)
Responsible Party: Sponsor-Investigator, Liming Cheng, Director, Head of orthopedics, Pricipal investigator, Clinical professor, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 56014768-4
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- with repair of deltoid ligament (Experimental): open reduction and internal fixation with repair of deltoid ligament
  Interventions: Procedure: repair of deltoid ligament
- without repair of deltoid ligament (No Intervention): open reduction and internal fixation without repair of deltoid ligament

INTERVENTIONS:
Procedure: repair of deltoid ligament — intraoperative repair of deltoid ligament combined with ORIF
  Arms: with repair of deltoid ligament

SUMMARY:
Ankle fracture is very common which is often combined with deltoid ligament injury. Although the incidence of deltoid ligament injury is high, but there is no unified and effective diagnosis method. Even whether the ankle fracture with deltoid ligament rupture needs surgical repair is still controversial. There is no high-level, multi-center, large sample, long-term follow-up clinical evidence to prove whether the repair of deltoid ligament is necessary or not. The main content of the project: 1 Achieve accurate classification of deltoid ligament rupture with intraoperative exploration. 2 Study the surgical indications and treatment guidelines by comparative study.

DETAILED DESCRIPTION:
Comparative study for ankle fracture combined with deltoid ligament rupture: with & without repair of ligament

ELIGIBILITY:
Inclusion Criteria:

* ankle fracture with deltoid ligament rupture

Exclusion Criteria:

* ankle fracture without deltoid ligament rupture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
AOFAS score | 12 months after surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fan J, Zhang X, Luo Y, You GW, Ng WK, Yang YF. Tibiotalocalcaneal (TTC) arthrodesis with reverse PHILOS plate and medial cannulated screws with lateral approach. BMC Musculoskelet Disord. 2017 Jul 24;18(1):317. doi: 10.1186/s12891-017-1666-2. PMID 28738797